CLINICAL TRIAL: NCT02380391
Title: EValuation of REsidual Platelet REactivity After Acute Coronary Syndrome in HIV-infected Patients. The EVERE2ST-HIV Study.
Brief Title: EValuation of REsidual Platelet REactivity After Acute Coronary Syndrome (ST+/ST-) in HIV
Acronym: EVERE2ST-HIV
Status: Completed | Type: Observational
Sponsor: Saint Antoine University Hospital (Other)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Franck Boccara, Professor of Cardiology, Saint Antoine University Hospital
Other Study IDs: EVERE2ST-HIV
Record Dates: First submitted 2015-02-24; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-02

CONDITIONS: Acute Coronary Syndrome; HIV
Keywords: Platelet reactivity; Acute coronary syndrome; Antiplatelet treatment; Antiretroviral treatment; HIV
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Each blood sample is composed of 5 tubes, for a total volume of 25 ml of blood :
  * 1 x 4.5 ml citrated tube : standard light transmission aggregometry
  * 1 x 4.5 ml citrated tube : Bedside test VerifyNow
  * 2 x 4.5 ml citrated tubes : flow cytometry
  * 1 x 7 ml EDTA tube : genetic analysis of cytochrome P450 2C19
  Blood samples do not require fasting.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- People living with HIV (HIV+): Adults experiencing first episode of ACS treated with percutaneous coronary intervention.
- People without HIV (HIV-): Adults experiencing first episode of ACS treated with percutaneous coronary intervention, matched to HIV+ on age, sex, known diabetes mellitus, and anti-platelet therapy.

SUMMARY:
Elevated on-treatment platelet reactivity is an independent risk factor of major adverse cardiovascular events following percutaneous coronary intervention or ACS. People living with HIV patients have a higher risk of recurrent events after ACS than people without HIV.

The investigators hypothesized that this increased risk is driven by higher platelet reactivity.

Using a nested case-control study design, HIV-infected and HIV-uninfected patients with a first episode of Acute Coronary Syndrome (ACS) treated with percutaneous coronary intervention were matched for age, sex, known diabetes mellitus and anti-platelet therapy.

The primary end-point was the residual platelet reactivity (RPA) on dual antiplatelet therapy assessed by light transmission aggregometry (LTA, 20µM ADP).

The study was conducted in a two large public university hospitals in central Paris, France.

DETAILED DESCRIPTION:
Study design :

Research of routine care - hospital based, two site, nested case-control study, conducted in the Institute of Cardiology within the Pitie-Salpetriere University Hospital and the Cardiac Center of the Saint Antoine University Hospital.

Number of participants :

Group 1 : n=80 HIV seropositive participants (HIV+) Group 2 : n=160 HIV seronegative participants (HIV-) Sample size calculation based on : 10% absolute difference between the two groups for maximum platelet aggregation (MPA) to residual platelet aggregation (RPA) ratio calculated MPA/RPA for each antiplatelet drug (Aspirin, Clopidogrel, Prasugrel).

Study justification :

Platelet function is a risk marker independent of ACS recurrence risk. People living with HIV who have a premature coronary artery disease, revealed by an ACS event, more frequently experience ischemic recurrence than people without HIV.

Hypothesis :

Due to their elevated residual platelet reactivity, people living with HIV present more frequent ACS recurrence following a first event than people without HIV.

Primary objective :

Determine if there is an influence of HIV and antiretroviral medications on the platelet reactivity of individuals under oral antiplatelet treatment. PLatelet reactivity will be assessed between one week to 3 years after the initial acute coronary syndrome under dual antiplatelet therapy.

Methods :

Platelet aggregation measured by :

1. Light transmission aggregometry (LTA, 20µM adenosine diphosphate receptor inhibitor (ADP) and 5µM of arachidonic acid (AA))
2. Point of care VerifyNowRM P2Y12 and ARU (P2Y12 Reaction Units and ARU Aspirin Reaction Units)
3. Flow cytometry (VAsodilatator Simulated Phosphoprotein (VASP))

ELIGIBILITY:
INCLUSION CRITERIA :

HIV+ group

* HIV-1 seropositive, known for a minimum of 6 months
* 18 years of age or older
* Hospitalisation for acute coronary syndrome a minimum of one month prior to inclusion (with or without coronary revascularisation)
* Under any antiplatelet therapy
* Willing and able to give informed consent to participate in the study

HIV- group

* HIV seronegative
* 18 years of age or older
* Hospitalisation for acute coronary syndrome a minimum of one month prior to inclusion (with or without coronary revascularisation)
* Under any antiplatelet therapy
* Willing and able to give informed consent to participate in the study

EXCLUSION CRITERIA :

* Refusal to give or sign informed consent
* Presence of a counterindication or non-indication for antiplatelet therapy
* Not associated with a social security regime (no health insurance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a history of acute coronary syndrome (at least one month before inclusion) with or without coronary revascularization and under any antiplatelet therapy.
  Controls matched on age (±5 years), sex, and known diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Residual platelet reactivity (measure 1). measured by light transmission aggregometry following stimulation by 20µM of ADP. | betwwen one week to 3 years
  Residual platelet reactivity under antiplatelet therapy measured by light transmission aggregometry following stimulation by 20µM of ADP.

SECONDARY OUTCOMES:
Residual platelet reactivity (measure 2). measured by light transmission aggregometry following stimulation by 5µM of arachidonic acid | betwwen one week to 3 years
  Residual platelet reactivity under aspirin measured by light transmission aggregometry following stimulation by 5µM of arachidonic acid.

CONTACTS AND LOCATIONS:
Overall Officials: Franck Boccara, MD, PhD, Principal Investigator — Saint Antoine University Hospital; Ariel Cohen, MD, PhD, Study Director — Saint Antoine University Hospital; Jean Philippe Collet, MD, PhD, Study Director — ACTION Study Group, Unité de Recherche Clinique-Hôpital Lariboisière (APHP) and Université Paris 6, INSERM, Paris, France; Johanne Silvain, MD, PhD, Study Director — ACTION Study Group, Unité de Recherche Clinique-Hôpital Lariboisière (APHP) and Université Paris 6, INSERM, Paris, France; Gilles Montalescot, MD, PhD, Study Chair — ACTION Study Group, Unité de Recherche Clinique-Hôpital Lariboisière (APHP) and Université Paris 6, INSERM, Paris, France
Locations (1):
- Cardiology department, Paris, France

REFERENCES:
- [Background] Parodi G, Marcucci R, Valenti R, Gori AM, Migliorini A, Giusti B, Buonamici P, Gensini GF, Abbate R, Antoniucci D. High residual platelet reactivity after clopidogrel loading and long-term cardiovascular events among patients with acute coronary syndromes undergoing PCI. JAMA. 2011 Sep 21;306(11):1215-23. doi: 10.1001/jama.2011.1332. PMID 21934054
- [Background] Boccara F, Mary-Krause M, Teiger E, Lang S, Lim P, Wahbi K, Beygui F, Milleron O, Gabriel Steg P, Funck-Brentano C, Slama M, Girard PM, Costagliola D, Cohen A; Prognosis of Acute Coronary Syndrome in HIV-infected patients (PACS) Investigators. Acute coronary syndrome in human immunodeficiency virus-infected patients: characteristics and 1 year prognosis. Eur Heart J. 2011 Jan;32(1):41-50. doi: 10.1093/eurheartj/ehq372. Epub 2010 Oct 21. PMID 20965887
- [Background] Lang S, Mary-Krause M, Cotte L, Gilquin J, Partisani M, Simon A, Boccara F, Bingham A, Costagliola D; French Hospital Database on HIV-ANRS CO4. Increased risk of myocardial infarction in HIV-infected patients in France, relative to the general population. AIDS. 2010 May 15;24(8):1228-30. doi: 10.1097/QAD.0b013e328339192f. PMID 20400883
- [Background] Triant VA, Lee H, Hadigan C, Grinspoon SK. Increased acute myocardial infarction rates and cardiovascular risk factors among patients with human immunodeficiency virus disease. J Clin Endocrinol Metab. 2007 Jul;92(7):2506-12. doi: 10.1210/jc.2006-2190. Epub 2007 Apr 24. PMID 17456578
- [Background] Friis-Moller N, Weber R, Reiss P, Thiebaut R, Kirk O, d'Arminio Monforte A, Pradier C, Morfeldt L, Mateu S, Law M, El-Sadr W, De Wit S, Sabin CA, Phillips AN, Lundgren JD; DAD study group. Cardiovascular disease risk factors in HIV patients--association with antiretroviral therapy. Results from the DAD study. AIDS. 2003 May 23;17(8):1179-93. doi: 10.1097/01.aids.0000060358.78202.c1. PMID 12819520
- [Background] Kaplan RC, Kingsley LA, Sharrett AR, Li X, Lazar J, Tien PC, Mack WJ, Cohen MH, Jacobson L, Gange SJ. Ten-year predicted coronary heart disease risk in HIV-infected men and women. Clin Infect Dis. 2007 Oct 15;45(8):1074-81. doi: 10.1086/521935. Epub 2007 Sep 12. PMID 17879928
- [Background] Patel P, Hanson DL, Sullivan PS, Novak RM, Moorman AC, Tong TC, Holmberg SD, Brooks JT; Adult and Adolescent Spectrum of Disease Project and HIV Outpatient Study Investigators. Incidence of types of cancer among HIV-infected persons compared with the general population in the United States, 1992-2003. Ann Intern Med. 2008 May 20;148(10):728-36. doi: 10.7326/0003-4819-148-10-200805200-00005. PMID 18490686
- [Background] Saves M, Chene G, Ducimetiere P, Leport C, Le Moal G, Amouyel P, Arveiler D, Ruidavets JB, Reynes J, Bingham A, Raffi F; French WHO MONICA Project and the APROCO (ANRS EP11) Study Group. Risk factors for coronary heart disease in patients treated for human immunodeficiency virus infection compared with the general population. Clin Infect Dis. 2003 Jul 15;37(2):292-8. doi: 10.1086/375844. Epub 2003 Jul 7. PMID 12856222
- [Background] Grinspoon SK. Metabolic syndrome and cardiovascular disease in patients with human immunodeficiency virus. Am J Med. 2005 Apr;118 Suppl 2:23S-28S. doi: 10.1016/j.amjmed.2005.01.047. PMID 15903292
- [Background] Capeau J. From lipodystrophy and insulin resistance to metabolic syndrome: HIV infection, treatment and aging. Curr Opin HIV AIDS. 2007 Jul;2(4):247-52. doi: 10.1097/COH.0b013e3281e66919. PMID 19372895
- [Background] Triant VA, Meigs JB, Grinspoon SK. Association of C-reactive protein and HIV infection with acute myocardial infarction. J Acquir Immune Defic Syndr. 2009 Jul 1;51(3):268-73. doi: 10.1097/QAI.0b013e3181a9992c. PMID 19387353
- [Background] Mangili A, Polak JF, Quach LA, Gerrior J, Wanke CA. Markers of atherosclerosis and inflammation and mortality in patients with HIV infection. Atherosclerosis. 2011 Feb;214(2):468-73. doi: 10.1016/j.atherosclerosis.2010.11.013. Epub 2010 Nov 17. PMID 21130995
- [Background] Coll B, Parra S, Alonso-Villaverde C, Aragones G, Montero M, Camps J, Joven J, Masana L. The role of immunity and inflammation in the progression of atherosclerosis in patients with HIV infection. Stroke. 2007 Sep;38(9):2477-84. doi: 10.1161/STROKEAHA.106.479030. Epub 2007 Aug 2. PMID 17673719
- [Background] Kaplan RC, Kingsley LA, Gange SJ, Benning L, Jacobson LP, Lazar J, Anastos K, Tien PC, Sharrett AR, Hodis HN. Low CD4+ T-cell count as a major atherosclerosis risk factor in HIV-infected women and men. AIDS. 2008 Aug 20;22(13):1615-24. doi: 10.1097/QAD.0b013e328300581d. PMID 18670221
- [Background] Torre D, Pugliese A. Platelets and HIV-1 infection: old and new aspects. Curr HIV Res. 2008 Sep;6(5):411-8. doi: 10.2174/157016208785861140. PMID 18855651
- [Background] Satchell CS, Cotter AG, O'Connor EF, Peace AJ, Tedesco AF, Clare A, Lambert JS, Sheehan GJ, Kenny D, Mallon PW. Platelet function and HIV: a case-control study. AIDS. 2010 Mar 13;24(5):649-57. doi: 10.1097/QAD.0b013e328336098c. PMID 20177361
- [Background] Boccara F, Mary-Krause M, Teiger E, et al. HIV-infected patients have an increased risk of recurrent ischemic events as compared to the general population after an acute coronary syndrome. Paper presented at: American Heart Association; November 15th, 2011, 2011; Orlando, USA.
- [Background] Baker JV, Neuhaus J, Duprez D, Kuller LH, Tracy R, Belloso WH, De Wit S, Drummond F, Lane HC, Ledergerber B, Lundgren J, Nixon DE, Paton NI, Neaton JD; INSIGHT SMART Study Group. Changes in inflammatory and coagulation biomarkers: a randomized comparison of immediate versus deferred antiretroviral therapy in patients with HIV infection. J Acquir Immune Defic Syndr. 2011 Jan 1;56(1):36-43. doi: 10.1097/QAI.0b013e3181f7f61a. PMID 20930640
- [Background] Scaradavou A. HIV-related thrombocytopenia. Blood Rev. 2002 Mar;16(1):73-6. doi: 10.1054/blre.2001.0188. PMID 11914001
- [Background] von Hentig N, Forster AK, Kuczka K, Klinkhardt U, Klauke S, Gute P, Staszewski S, Harder S, Graff J. Platelet-leucocyte adhesion markers before and after the initiation of antiretroviral therapy with HIV protease inhibitors. J Antimicrob Chemother. 2008 Nov;62(5):1118-21. doi: 10.1093/jac/dkn333. Epub 2008 Aug 27. PMID 18753189
- [Background] Corrales-Medina VF, Simkins J, Chirinos JA, Serpa JA, Horstman LL, Jy W, Ahn YS. Increased levels of platelet microparticles in HIV-infected patients with good response to highly active antiretroviral therapy. J Acquir Immune Defic Syndr. 2010 Jun;54(2):217-8. doi: 10.1097/QAI.0b013e3181c8f4c9. No abstract available. PMID 20505474
- [Background] Baker J, Ayenew W, Quick H, Hullsiek KH, Tracy R, Henry K, Duprez D, Neaton JD. High-density lipoprotein particles and markers of inflammation and thrombotic activity in patients with untreated HIV infection. J Infect Dis. 2010 Jan 15;201(2):285-92. doi: 10.1086/649560. PMID 19954384
- [Background] Daali Y, Ancrenaz V, Bosilkovska M, Dayer P, Desmeules J. Ritonavir inhibits the two main prasugrel bioactivation pathways in vitro: a potential drug-drug interaction in HIV patients. Metabolism. 2011 Nov;60(11):1584-9. doi: 10.1016/j.metabol.2011.03.015. Epub 2011 May 6. PMID 21550074
- [Background] Collet JP, Cayla G, Cuisset T, Elhadad S, Range G, Vicaut E, Montalescot G. Randomized comparison of platelet function monitoring to adjust antiplatelet therapy versus standard of care: rationale and design of the assessment with a double randomization of (1) a fixed dose versus a monitoring-guided dose of aspirin and clopidogrel after DES implantation, and (2) treatment interruption versus continuation, 1 year after stenting (ARCTIC) study. Am Heart J. 2011 Jan;161(1):5-12.e5. doi: 10.1016/j.ahj.2010.09.029. PMID 21167334
- [Background] Silvain J, Bellemain-Appaix A, Barthelemy O, Beygui F, Collet JP, Montalescot G. Optimal use of thienopyridines in non-ST-elevation acute coronary syndrome following CURRENT-OASIS 7. Circ Cardiovasc Interv. 2011 Feb 1;4(1):95-103. doi: 10.1161/CIRCINTERVENTIONS.109.910406. No abstract available. PMID 21325198
- [Background] Silvain J, Collet JP, Nagaswami C, Beygui F, Edmondson KE, Bellemain-Appaix A, Cayla G, Pena A, Brugier D, Barthelemy O, Montalescot G, Weisel JW. Composition of coronary thrombus in acute myocardial infarction. J Am Coll Cardiol. 2011 Mar 22;57(12):1359-67. doi: 10.1016/j.jacc.2010.09.077. PMID 21414532
- [Background] Hulot JS, Collet JP, Cayla G, Silvain J, Allanic F, Bellemain-Appaix A, Scott SA, Montalescot G. CYP2C19 but not PON1 genetic variants influence clopidogrel pharmacokinetics, pharmacodynamics, and clinical efficacy in post-myocardial infarction patients. Circ Cardiovasc Interv. 2011 Oct 1;4(5):422-8. doi: 10.1161/CIRCINTERVENTIONS.111.963025. Epub 2011 Oct 4. PMID 21972404
- [Background] Silvain J, Cayla G, Hulot JS, Finzi J, Kerneis M, O'Connor SA, Bellemain-Appaix A, Barthelemy O, Beygui F, Collet JP, Montalescot G. High on-thienopyridine platelet reactivity in elderly coronary patients: the SENIOR-PLATELET study. Eur Heart J. 2012 May;33(10):1241-9. doi: 10.1093/eurheartj/ehr407. Epub 2011 Nov 7. PMID 22067090